CLINICAL TRIAL: NCT05805904
Title: A Double-blind, Placebo-controlled, Randomized, Single and Multiple Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986278 in Healthy Chinese Participants
Brief Title: A Study to Evaluate the Drug Levels, Safety, and Tolerability of BMS-986278 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM027-067
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: BMS-986278; Drug: Placebo
- Group 2 (Experimental)
  Interventions: Drug: BMS-986278; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days.
Drug: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the drug levels, safety, and tolerability of BMS-986278 in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Chinese (both biological parents are ethnically Chinese).
* Healthy Chinese male and female (women not of child bearing potential) participants as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECGs, or clinical laboratory determinations.
* Body mass index of 18.0 to 28.0 kg/m2, inclusive. Body mass index = weight (kg)/(height [m])2.
* Body weight ≥ 50 kg

Exclusion Criteria:

* Any significant acute or chronic medical illness that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* Current or recent (within 3 months of study intervention administration) gastrointestinal (GI) disease that could affect the absorption, distribution, metabolism, and excretion of study drug (eg, bariatric procedure, Gilbert's syndrome)
* Any GI surgery (eg, cholecystectomy and any other GI surgery) that, in the opinion of the investigator, could impact the absorption of study treatment (uncomplicated appendectomy and hernia repair are acceptable)
* Women who are of childbearing potential
* Women who are breastfeeding
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory determinations beyond what is consistent with the target population. Have abnormal renal function at screening, as evidenced by an estimated glomerular filtration rate < 90 mL/min/1.732 m^2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula and the absence of protein in urine

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 19
Time of maximum observed concentration (Tmax) | Up to Day 19
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 19

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 26
Number of participants with physical examination abnormalities | Up to Day 19
Number of participants with vital sign abnormalities | Up to Day 19
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 19
Number of participants with clinical laboratory abnormalities | Up to Day 19
Cmax | Up to Day 19
Tmax | Up to Day 19
AUC(0-T) | Up to Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Shanghai, China

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm